CLINICAL TRIAL: NCT04501523
Title: A Prospective, Phase II Trial Using Circulating Tumor DNA to Initiate Post-operation Boost Therapy After Neoadjuvant Chemotherapy in Triple-negative Breast Cancer
Brief Title: A Prospective, Phase II Trial Using ctDNA to Initiate Post-operation Boost Therapy After NAC in TNBC
Acronym: Apollo
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liu Qiang, Doctor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SunYatsenU2H-LQ3
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — tislelizumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A (Experimental): ctDNA positive, non-pCR Intervention: Tislelizumab(anti-PD1 antibody) combined with capecitabine
  Interventions: Drug: Tislelizumab; Drug: capecitabine
- B (Active Comparator): ctDNA positive, non-pCR Intervention: capecitabine(standard care)
  Interventions: Drug: capecitabine
- C (Experimental): ctDNA positive, pCR Intervention: capecitabine
  Interventions: Drug: capecitabine
- D (No Intervention): Follow up(standard care)

INTERVENTIONS:
Drug: Tislelizumab — 200mg, q3w, for 1 year
  Arms: A
Drug: capecitabine — 600-750 mg/m2 PO Bid，continuous, for 1 year
  Arms: A; B; C

SUMMARY:
Positive circulating tumor DNA(ctDNA) status is associated with worse prognosis in breast cancer, especially triple-negative breast cancer(TNBC). Our trial aims to improve the outcome of TNBC patients by using ctDNA to identify patients with high relapse risk. ctDNA positive patients will be randomized to receive boost therapy or standard therapy indicated in NCCN guidelines after NAC.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed triple negative (ER-/PR-/HER2-) invasive breast cancer, clinical stage II-III at diagnosis (AJCC 6th edition) based on initial evaluation by physical examination and/or breast imaging prior to study registration.ER and PR will be considered negative if ≤ 1% of cells stain weakly positive. HER2 will be considered negative if scored 0 or 1+ by immunohistochemistry (IHC) or 2+ by IHC associated with a fluorescence in situ hybridization (FISH) ratio of < 2.0 or < 6 copies per cell.
* Must receive preoperative (neoadjuvant) chemotherapy. NOTE: Acceptable preoperative regimens include those recommended by NCCN guidelines. Participants who received preoperative therapy as part of a clinical trial may enroll.
* ctDNA positive at baseline, after NAC or after surgery
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Written informed consent to provide research blood samples and tumor samples
* Patients must be willing to have frequent blood tests (every 3 months ) and receive a 12 month course of tislelizumab if randomised to tislelizumab treatment on ctDNA detection
* No evidence of distant metastatic disease on staging scans conducted at the time of diagnosis

Exclusion Criteria:

* Previously participated in other interventional trials
* Previous malignancy within 3 years of breast cancer diagnosis
* Pregnancy or breastfeeding
* No written consent
* Unable to receive standard NAC and subsequent radiotherapy(if needed)
* Active autoimmune disease

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
5 years Disease free survival(DFS) | 60 months
  From diagnosis to 5yrs or DFS events; To determine 5-year disease free survival in ctDNA positive participants with confirmed triple negative breast cancer (TNBC) treated with a boost therapy or standard of care following preoperative chemotherapy

SECONDARY OUTCOMES:
5 years overall survival(OS) | 60 months
  From diagnosis to 5yrs or death; To determine 5-year overall survival in ctDNA positive participants with confirmed triple negative breast cancer (TNBC) treated with a boost therapy or standard of care following preoperative chemotherapy
pathological complete remission(pCR) rate | 12 months
  pathological complete remission
brain metastasis rate | 60 months
  The percentage of patients who develop brain metastasis
objective response rate(ORR) | 12 months
  The percentage of patients who achieved PR+CR
Number of Patients with Adverse Events as a Measure of Safety and Tolerability | 12 months
  To determine the toxicities associated with tislelizumab in this population
10 years DFS | 120 months
  To determine 10-year disease free survival in ctDNA positive participants with confirmed triple negative breast cancer (TNBC) treated with a boost therapy or standard of care following preoperative chemotherapy
10 years OS | 120 months
  To determine 10-year overall survival in ctDNA positive participants with confirmed triple negative breast cancer (TNBC) treated with a boost therapy or standard of care following preoperative chemotherapy
Relapse and metastasis rate | 24 months
  The percentage of patients who develop brain metastasis any relapse or metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Liu, MD, Principal Investigator — Sunyat-sen Memorial Hospital
Locations (1):
- Sunyat-sen Memorial Hospital, Guandong, Guangdong, China